CLINICAL TRIAL: NCT06133426
Title: Evaluation of the Role of Connected Scales in the Therapeutic Care of Hematology Patients
Acronym: BTP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Withings (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: APHP230916; 2023-A01684-41 (Other: IDRCB)
Record Dates: First submitted 2023-10-30; First posted 2023-11-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Lymphoma, Non-Hodgkin; Myeloma Multiple
Keywords: Hematology; Connected scale; Remote monitoring
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Pilot study of feasibility and acceptability, non-comparative, non-controlled, non-randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort group (Other): Patients will be used a connected scale during the duration of their participation in the study.
  Patients will be invited to use the scale once a day. Patient's data will be accesible by medical team via a specific remote plateform.
  Alert will be generated according to the evolution of clinical data, permetting a early patient management by the medical team.
  Interventions: Device: Connected scale "Body Comp Pro" from Withings

INTERVENTIONS:
Device: Connected scale "Body Comp Pro" from Withings — Use once a day from inclusion to week 7.

SUMMARY:
In this research, we will evaluate the feasibility of following by remote monitoring, using a connected scale, in hematology patients suffering from myeloma or lymphoma and requiring treatment with chemotherapy. 30 patients will be included in the research and will all use a connected scale for the duration of their participation (7 weeks +/- 1 week). During their participation, patients will be asked to weigh themselves once a day, ideally at a set time. Patient data will be accessible by the medical team via a remote monitoring platform.

Alerts will be generated in the event of abnormal development of certain clinical parameters (weight, heart rate, etc.) allowing early treatment to be implemented by the medical team.

At the end of their participation, we will evaluate patients' support and perception of this tool, as well as the healthcare consequences of the alerts generated by the remote monitoring platform.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 and over (male or female)
* Patient suffering from aggressive non-Hodgkin's lymphoma or multiple myeloma with a plan for systemic chemotherapy or having started two cycles or less or patient with the need for therapeutic intensification under the cover of autograft in the context of myeloma or lymphoma
* Patient who can be contacted by telephone during their participation in the research
* Patient able to return home at the end of their initial hospitalization
* Patient affiliated to social security
* Patient able to read and speak French
* Patient having signed free, informed and written consent

Exclusion Criteria:

* Patient with an estimated life expectancy < 3 months
* Patient with moderate to severe cognitive impairment (assessed by MMSE < 20)
* Patient with a psychiatric or physical disability that does not allow the use of the device
* Patient with a pacemaker
* Patient participating in another intervention research project
* Pregnant patient
* Patient deprived of liberty
* Patient under legal protection (guardianship or curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who agreed to participate in research | Inclusion
  Number of included patients / Number of indormed patients

SECONDARY OUTCOMES:
Frequency of use of the connected scale during the patient's participation in the research | From inclusion to week 7
  Average of weighings/week
Assessment of the patient's anxiety regarding the device | week 7
  Specific 5 points Likert Scale (1 - 5 ; Higher score mean a worse outcome)
Evaluation of the ease of use of the device perceived by the patient | week 7
  Symptom Usability Scale (0 - 100 ; Higher score mean a better outcome)
Evaluation of the implementation of the study by the patient | week 7
  FIM (Feasibility of Intervention Measure), AIM (Acceptability of Intervention Measure) and IAM (Intervention Appropriateness Measure) / (1 - 5 ; Higher score mean a better outcome)
Evaluation of the consequences in care of alerts generated by the plateform | From inclusion to week 7
  Number of alerts generated/patient.
Evaluation of the consequences in care of alerts generated by the plateform | From inclusion to week 7
  Number of calls made/patient.
Evaluation of the consequences in care of alerts generated by the plateform | From inclusion to week 7
  Average time spent per call following the generation of an alert.
Evaluation of the consequences in care of alerts generated by the plateform | From inclusion to week 7
  Number and type of consultations, hospitalizations, additional assessments resulting from the generation of an alert.

CONTACTS AND LOCATIONS:
Locations (1):
- Cochin Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No